CLINICAL TRIAL: NCT01182025
Title: A Clinical Trial to Evaluate the Effectiveness and Safety of Xiyanping Injection in the Treatment of Mild Type of Hand, Foot, and Mouth Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Collaborators: Beijing University of Chinese Medicine (Other); China Academy of Chinese Medical Sciences (Other)
Responsible Party: Guoliang Zhang, The First Affiliated Hospital of Anhui College of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200907001-4
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Mild type of hand, foot and mouth disease; Xiyanping Injection; Effectiveness; Safety
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Mouth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Western therapy (Active Comparator)
  Interventions: Other: Western therapy
- Xiyanping Injection (Experimental)
  Interventions: Drug: Xiyanping Injection
- Xiyanping Injection with western medicine (Experimental)
  Interventions: Drug: Xiyanping Injection with western medicine

INTERVENTIONS:
Other: Western therapy — Symptomatic treatment: vitamin B, vitamin C, mouth care and skin care.
  1. Adopting physical cooling therapy, including physical cooling paste or warm bathing, when patient's body temperature is lower than 38.5 degree Celsius;
  2. Using Ibuprofen suspension when patient's temperature higher than 38.5 degree Celsius;
  Arms: Western therapy
Drug: Xiyanping Injection — Dosage for child medication:
  5-10mg/kg/d (0.2-0.4ml/kg/d) in 5% Glucose solution, IV, with speed of 20-30 drops per minute, each day; or as directed by doctor.
  Arms: Xiyanping Injection
Drug: Xiyanping Injection with western medicine — 1. Symptomatic treatment using the same treatment methods in western therapy group;
  2. Symptomatic treatment using the same treatment methods in Xiyanpin injection group.
  Arms: Xiyanping Injection with western medicine

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of Xiyanping Injection for mild type of hand, foot, and mouth disease.

DETAILED DESCRIPTION:
By adopting a multi-center, randomized and controlled clinical trial, this study is aimed to evaluate the efficacy and safety of Xiyanping Injection in the treatment of mild type of Hand, Foot and Mouth Disease (HFMD), and designed to combine both observational and interventional methodologies in this research.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe hand-foot-mouth disease patients according to Hand-Foot-Mouth Disease Treatment Guidelines 2010 issued by China's Ministry of Health; More than 1/3 patients should be diagnosed by etiological examination.
* Less than 48 hours of occurrence of fever and/or occurrence of tetter or herpes.
* Age of 1-14 years.
* Patients or their guardians agree to participate in this study and signed the informed consent form.

Exclusion Criteria:

* Complicated with other serious primary diseases in organ such as congenital heart disease, chronic hepatitis, nephritis and blood diseases, etc.
* With history of allergies on traditional Chinese medicine.
* Patients or their guardians suffering from Psychiatric diseases.
* Attending other clinical studies on HFMD after diagnosed.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-05 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
time of bringing down the fever | 10 days
  Refering to the length of time to bring down the fever by 0.5 degrees Celsius after the medicine is taken.
time of body temperature going back to normal | 10 days
  Refering to the time of the armpit temperature of lower than 37.0 degrees Celsius, lasting for at least 24 hours, after the medicine is taken.

SECONDARY OUTCOMES:
time of symptom disappearance | 10 days
  Refering to the length of time when clinical symptoms and signs totally disappere after the medicine is used.
case severity rate | 10 days
  Refering to the ratio of patient with mild type of HFMD to severe type, such as damage of central nervous system, pulmonary edema, heart failure, respiratory failure, etc.
time of tetter disappearance | 10 days
  Refering to the length of time when the tetter due to HFMD disappears, characterised by scab(s) or dropping; and time of oral ulcer concrescence, etc.
direct medical cost | 10 days
  Referring to the costs in the treatment of HFMD and relative disease, including the registration fee, examination fee, and drug fees, etc.
safety outcome | 10 days
  Calculated by adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Zhang, Principal Investigator — An'Hui Chinese Medical College Affiliated No.1 Hospital
Locations (5):
- China (5):
  - Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Shenzhen Maternity & Child Healthcare Hospital, Shenzhen, Guangzhou
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi